CLINICAL TRIAL: NCT01639196
Title: The Expressive Writing Paradigm: A Study of Therapeutic Effectiveness for Chronic Pain
Brief Title: Brief Online Intervention for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 338877-1
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Psychological adjustment; Writing; Brief intervention; Online; Internet interventions
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-compassion writing (Experimental)
  Interventions: Other: Self-compassion writing
- Self-efficacy writing (Active Comparator)
  Interventions: Other: Self-efficacy writing

INTERVENTIONS:
Other: Self-compassion writing — Participants are instructed to write about their chronic pain in a way that elicits self-compassion for 20 minutes once a week for three consecutive weeks.
  Arms: Self-compassion writing
Other: Self-efficacy writing — Participants are instructed to write about their chronic pain in a way that elicits self-efficacy for 20 minutes once a week for three consecutive weeks.
  Arms: Self-efficacy writing

SUMMARY:
The purpose of this study is to explore the effects of writing about chronic pain on mental and physical health. The effectiveness of two different types of brief online writing interventions will be explored in individuals with chronic pain.

DETAILED DESCRIPTION:
Chronic pain is highly prevalent and costly, but often not treated effectively. Psychological interventions are needed as part of chronic pain treatment since the pain affects many aspects of an individual's life. In particular, brief psychological interventions that are easily accessible (i.e., online) could benefit many people with chronic pain. Writing interventions have been used in recent years to understand difficult experiences. Writing interventions have been found to help individuals explore distressing thoughts and feelings, such as those that are associated with pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic pain or a chronic pain condition or discussed pain management strategies (e.g., pain medication) with a doctor
* Experience pain on most days of the month for at least six months
* Able to read and write in English

Exclusion Criteria:

* Chronic pain directly caused by a terminal condition (e.g., stage 4 cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Compassion Scale | Change from Baseline in Self-Compassion Scale at 4 weeks
Change from Baseline in Pain Self-Efficacy Scale | Change from Baseline in Pain Self-Efficacy Scale at 4 weeks

SECONDARY OUTCOMES:
Change from Baseline in Pain Severity | Change from Baseline in Pain Severity at 4 weeks
  Pain severity is measured on a 10-point rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Hoffman, PhD, Principal Investigator — University of Maryland, College Park